CLINICAL TRIAL: NCT05598801
Title: A Single-center, Prospective, Clinical Study of VersaWrap Utilization in the Hand
Status: Completed | Type: Observational
Sponsor: Research Source (Network)
Responsible Party: Sponsor
Other Study IDs: VW-001- Version 02
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Tendon Repair; Fracture Repair; Tenolysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- VersaWrap: All enrolled patients will received VersaWrap applied prior to surgical closure on the affected tendon.
  Interventions: Device: VersaWrap

INTERVENTIONS:
Device: VersaWrap — VersaWrap is applied to the affected tendon to allow post-operative gliding.

SUMMARY:
The purpose of this study is to evaluate the efficacy on the use of VersaWrap® in surgery of the hand/fingers, including tendon repair, fracture repair, or tenolysis of the hand/fingers. VersaWrap is designed to allow tendon gliding and to protect tendon gliding postoperatively

DETAILED DESCRIPTION:
This is a prospective, post-market, observational, single center study evaluating the use of VersaWrap. Patients identified by the Investigator in his practice as needing surgery of the hand/fingers and meeting all the inclusion and none of the exclusion. Patients will consent to participating in the study, prior to any study procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-70 at the time of surgery
2. Patients undergoing hand/finger surgery, including tendon repair, fracture repair or tenolysis
3. Psychosocially, mentally and physically able to fully comply with this protocol including adhering to follow-up schedule, study requirements with a signed informed consent with a study collaborator present at the time of signing to ensure compliance.

Exclusion Criteria:

1. Non-English speaking
2. Known allergy or sensitivity to citrate, alginate or hyaluronate
3. Pregnant or breastfeeding
4. Currently a prisoner
5. Patient has any condition, that in the opinion of the Investigator, would prohibit the patient from complying with the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who meet the following inclusion criteria and none of the exclusion criteria will be enrolled in the study. A patient is considered enrolled upon placement of the VersaWrap during the surgical procedure. If the surgeon decides intra-operatively not to utilize the VersaWrap, the patient will be considered a screen failure.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-08-17 (Actual); Study Completion 2025-08-17 (Actual)

PRIMARY OUTCOMES:
Number of participants diagnosed with post-operative tenolysis | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Austin Hand Group, Austin, Texas, United States